CLINICAL TRIAL: NCT02820103
Title: Reducing Patient Delay in Acute Coronary Syndrome (RAPiD): A Web-based Randomised Controlled Trial Examining the Effect of a Behaviour Change Intervention on Participants' Intentions to Seek Help
Brief Title: Reducing Acute Coronary Syndrome Patient Delay
Acronym: RAPiD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Edinburgh Napier University (Other)
Collaborators: University of Stirling (Other); University of Aberdeen (Other); University of Dundee (Other); The University of New South Wales (Other)
Responsible Party: Principal Investigator, Barbara Farquharson, Dr Barbara Farquharson, Edinburgh Napier University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: CZH/4/1025
Record Dates: First submitted 2016-06-21; First posted 2016-06-30 (Estimated); Last update posted 2017-08-16 (Actual); Status verified 2017-08

CONDITIONS: Acute Coronary Syndrome
Keywords: Patient delay; Behaviour change; Intervention Modelling Experiment
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Information leaflet (control) (Active Comparator): Participants in the control group will receive information that is currently used routinely in the NHS site to inform patients with ACS what to do if they experience symptoms after discharge. The information from two leaflets: 1. 'Using GTN', produced by the hospital and 'Angina' produced by the British Heart Foundation, published 08/04/2014 and available at https://www.bhf.org.uk/publications/heart-conditions/angina . The information explains the symptoms of angina and heart attack and advises what to do in the event of experiencing these symptoms. This information will be presented in written text format on screen.
  Interventions: Behavioral: Leaflet information (control)
- Text+Visual BCT-based intervention (Intervention Group 1) (Experimental): Participants in the visual intervention group will receive the control condition specified above PLUS a specifically developed Text+Visual BCT-based intervention, comprising the 12 BCTs identified earlier in a Systematic Review and expert consensus study. The BCTs are Problem solving; Action planning; Social support (practical); Social support (emotional); Instruction on how to perform the behaviour; Information about health consequences; Salience of health consequences; Prompts/cues; Credible source; Pro's & Con's; Comparative imagining of future outcomes; Mental rehearsal of successful performance
  Interventions: Behavioral: Text+Visual BCT-based intervention; Behavioral: Leaflet information (control)
- Text-only BCT-based intervention (Intervention Group 2) (Experimental): Information leaflet (usual care) plus text-only BCT-based intervention (Intervention group 2) Participants in the text-only BCT-based intervention group will receive the control condition specified above plus a text-only BCT-based intervention. This was developed in the same way as the text+visual BCT-based intervention but does not include the visual elements (i.e. animation). Instead, the voiceover from the animated film is displayed in text on screen instead.
  Interventions: Behavioral: Text-only BCT intervention; Behavioral: Leaflet information (control)

INTERVENTIONS:
Behavioral: Text+Visual BCT-based intervention — Participants in the visual intervention group will receive usual care specified below plus a specifically developed Text + Visual BCT-based intervention, comprising 12 BCTs identified from SR and expert consensus study. An animated video, just under 8 minutes in length is hosted online in the Intervention Modelling Experiment. The animation contains 9 of the 12 BCTs and tells the 'delay stories' of three different characters. It was not possible to deliver all of the 12 BCTs comprehensively in the relatively passive media of the animation as some techniques require active participation from participants (e.g. action planning). Thus, n=7 BCTs (1 2 Problem-solving; 1 4 Action planning; 5 2 Salience of consequences; 7 1 Prompts/cues; 9 3 Comparative imagining of future outcomes; 15 2 Mental rehearsal of successful performance) are also delivered via short web-based exercises which follow the animation.
  Arms: Text+Visual BCT-based intervention (Intervention Group 1)
Behavioral: Text-only BCT intervention — Participants in the text-only BCT-based intervention group will receive the usual care specified above plus a text-only BCT-based intervention. This was developed in the same way as the text + visual BCT-based intervention but does not include the visual elements (i.e. animation). Instead, the voiceover from the animated film is displayed in text on screen and narrated in audio. The BCTs which require active engagement are delivered via identical web-based exercises as the text + visual BCT-based intervention.
  Arms: Text-only BCT-based intervention (Intervention Group 2)
Behavioral: Leaflet information (control) — Participants in the control group will receive information that is currently used routinely in the NHS site to inform patients with ACS what to do if they experience symptoms after discharge.

SUMMARY:
1. To test the effectiveness of the theory-based interventions (text+visual and text-only BCT-based interventions) against usual care in changing patients' intentions to phone ambulance immediately with symptoms of ACS ≥ 15 minutes duration.
2. To determine the most effective mode of delivery by comparing the text+visual BCT-based intervention with text-only BCT-based intervention.
3. To investigate any unintended consequences of the intervention on intentions to phone an ambulance for non-life-threatening symptoms.

DETAILED DESCRIPTION:
Patient delay means many people do not achieve optimal benefit of time-dependent treatments for Acute Coronary Syndrome (ACS). Reducing delay would reduce mortality and morbidity but to date, interventions to change behaviour have had mixed results. Systematic inclusion of behaviour-change techniques (BCTs) or a visual mode of delivery might improve the efficacy of interventions.

Aim To evaluate the efficacy of a BCT-based intervention and to compare two possible modes of delivery (text+visual and text-only).

Design A 3-arm web-based, parallel randomised, controlled trial of a theory-based intervention.

Methods and analysis The intervention comprises 12 BCTs systematically identified following systematic review and a consensus exercise undertaken with behaviour change experts. We aim to recruit n=177 participants who have experienced ACS in the previous 6 months from a local National Health Service (NHS) Teaching Hospital. Participants will be identified by Cardiac Rehabilitation staff and invited by letter to take part in the study. Those who wish to take part will be asked to access the experiment at a secure web-address and consent re-checked. Consenting participants will be randomly allocated in equal numbers to one of three study groups: i) usual care ii) usual care plus text-only BCT-based intervention or iii) usual care plus text+visual BCT-based intervention. The outcome variable will be the change in intention to phone an ambulance immediately with symptoms of ACS ≥15 minutes duration assessed using two randomised series of 8 scenarios representing varied symptoms before and after delivery of the interventions or control condition (usual care).

ELIGIBILITY:
Inclusion Criteria:

* Adults, aged > 18 years
* Experience of Acute Coronary Syndrome within the previous six months

Exclusion Criteria:

* Anyone still hospitalised
* People who have experienced ACS within the previous two weeks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 177 (Estimated)
Dates: Start 2017-02-20 (Actual); Primary Completion 2017-10 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
Intentions to phone an ambulance immediately in response to scenarios representing possible symptoms of ACS using a 7-point Likert scale. | Immediately post intervention
  Intention: Informed by the Theory of Planned Behaviour (Ajzen 1991), participants' intentions to phone an ambulance immediately will be assessed in response to each scenario using a single Likert-type item ('For these symptoms, after this amount of time, I would phone an ambulance immediately') scored 1=strongly disagree to 7=strongly agree.

SECONDARY OUTCOMES:
Illness and symptom perceptions measured using the brief Illness Perception Questionnaire | Immediately post intervention
  Participants' illness representations in relation to symptoms presented in each scenario will be assessed using the Brief Illness Perception Questionnaire (B-IPQ) (Broadbent et al. 2006). The questionnaire consists of 9 items assessing the five components that make up a person's perception of their illness - identity (beliefs about the illness label and symptoms), cause (beliefs about factors responsible for causing illness), timeline (beliefs and expectations about the course of illness), consequences (beliefs and expectations about the impact of illness) and cure-control (beliefs about the efficacy of treatment or coping behaviours). The questionnaire has good test-retest reliability, has been validated among people with Myocardial Infarction (MI) and has been shown able to distinguish between different illnesses (Broadbent et al. 2006).
Cognitive determinants of intention assessed using questionnaire based upon the theory of planned behaviour. | Immediately post intervention
  : Informed by the Theory of Planned Behaviour (Ajzen 1991), the questionnaire will include - three items assessing attitude toward phoning an ambulance immediately using semantic differential scales (e.g. Useless-Useful) scored 1 to 7; three subjective norm items (e.g. people who are important to me think I should phone ambulance immediately in this situation) scored 1=Strongly disagree to 7=Strongly agree; and three perceived behavioural control items (e.g. Phoning an ambulance immediately in this situation is beyond my control) scored 1=Strongly disagree to 7=Strongly agree.
Self-efficacy assessed using questionnaire based upon Social Cognitive theory | Immediately post intervention
  Informed by the Social Cognitive Model (Bandura 1998), people's generic self-efficacy to call an ambulance immediately will be assessed once before and once after the intervention. Participants will be asked to rate how certain they are that they could phone an ambulance immediately in nine different situations which vary in how difficult it would be to phone an ambulance (e.g. if you were out with friends). Responses will be elicited on a scale ranging from 0=not at all certain to 100=highly certain.

CONTACTS AND LOCATIONS:
Locations (1):
- NHS Tayside, Dundee, Tayside, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Farquharson B, Dombrowski S, Pollock A, Johnston M, Treweek S, Williams B, Smith K, Dougall N, Jones C, Pringle S. Reducing patient delay with symptoms of acute coronary syndrome: a research protocol for a systematic review of previous interventions to investigate which behaviour change techniques are associated with effective interventions. Open Heart. 2014 Aug 12;1(1):e000079. doi: 10.1136/openhrt-2014-000079. eCollection 2014. PMID 25332805
- [Derived] Farquharson B, Johnston M, Williams B, Smith K, Dombrowski S, Jones C, Treweek S, Dougall N, Grindle M, Savinc J, Abyhankar P. Reducing patient delay in acute coronary syndrome: Randomized controlled trial testing effect of behaviour change intervention on intentions to seek help. Br J Health Psychol. 2023 Feb;28(1):188-207. doi: 10.1111/bjhp.12619. Epub 2022 Aug 8. PMID 35942523
- [Derived] Farquharson B, Johnston M, Smith K, Williams B, Treweek S, Dombrowski SU, Dougall N, Abhyankar P, Grindle M. Reducing patient delay in Acute Coronary Syndrome (RAPiD): research protocol for a web-based randomized controlled trial examining the effect of a behaviour change intervention. J Adv Nurs. 2017 May;73(5):1220-1234. doi: 10.1111/jan.13191. Epub 2016 Nov 18. PMID 27779777